CLINICAL TRIAL: NCT03221361
Title: Maximum Biting Force of Injectable Thermoplastic Resin Versus Conventional Resin in Complete Denture Patients (A Randomized Clinical Trial)
Brief Title: Maximum Biting Force of Inject Able Thermoplastic Resin Versus Conventional Resin in Complete Denture Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed saad eid, Dr., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 28711170100211
Record Dates: First submitted 2017-07-16; First posted 2017-07-18 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Biting Force

STUDY DESIGN:
Intervention Model Description: prospective , parallel , randomized clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The study will be blinded regarding the statistician who is responsible for data analysis.
  The participant patients will be blinded. The outcome assessor for biting force can be blinded during the measurement, the operator cannot be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoplastic resin group (Active Comparator): Thermoplastic complete denture placement is done
  Interventions: Device: thermoplastic complete denture
- conventional acrylic resin group (Placebo Comparator): conventional acrylic resin complete denture placement is done
  Interventions: Device: conventional acrylic resin complete denture

INTERVENTIONS:
Device: thermoplastic complete denture — a device used ti substitute teeth for edentlous patient made of thermoplastic resin
  Arms: Thermoplastic resin group
Device: conventional acrylic resin complete denture — A device used to substitute the teeth for edentlous patient made of acrylic resin
  Arms: conventional acrylic resin group

SUMMARY:
In this research we are comparing the new thermoplastic material side by side with the conventional poly methyl methacrylate for fully edentulous patients measuring their maximum biting force whether it is going to be higher by the new polyamide material.

DETAILED DESCRIPTION:
For all included patients and in the first visit, panoramic x ray is taken then a primary impression will be made for the maxillary and mandibular arches using irreversible hydrocolloid material. Then, the maxillary and mandibular impressions will be poured with a hard stone to get a study casts.

A double layer wax spaced self-cured acrylic resin will be used to prepare a special tray for each patient. The special tray using also irreversible hydrocolloid material makes a secondary impression. The secondary impressions will be poured using extra hard dental stone to get the master casts.

At this point the patient is given a number to enter one of the two groups either the intervention group or the control group.

For the intervention group, the framework of the thermoplastic resin is usually thicker than that of the metal. At this time the framework wax pattern will be ready for spruing and flasking using specially designed flasks. The injection of the thermoplastic resin will be started after the elimination of wax and the procedure will be done using thermopress machine.

In the third visit for all patients, the finished denture bases of thermoplastic resin will be tried inside the patient's mouth to check its fitting, retention, reciprocation and opposing occlusion.

Then, a face bow record will be taken for each patient which will be used to mount the maxillary cast on the articulator. For mounting the mandibular cast, either an intercuspal or centric jaw relation will be used. Artificial teeth will be set up and tried in in the patient's mouth in the fourth visit to check esthetics, phonetics, lip support, occlusion and uneven pairing.

In The fifth visit, the finished prosthesis will be adjusted and delivered to each patient, the outcome data will be collected using a questionnaire, and a salivary swap is taken for microbial count detection.

Complete dentures will be constructed for all patients; Group- I: patients will receive complete dentures from thermoplastic material Group- II: patients will receive complete dentures from conventional Poly methyl Methacrelate resin.

Then use Gnatho-dynamometer for measure the biting force for all patients

ELIGIBILITY:
Inclusion Criteria:

* - Completely edentulous
* No bone irregularities
* Good oral hygiene
* Should be co-operative
* Medically free
* No TMJ Problems

Exclusion Criteria:

* - Bone irregularities , soft tissue ulcerations , severe undercuts
* Serious systemic problem
* Patient with xerostomia
* Severely resorbed ridge

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
maximum biting force | 0,2,4,6 months
  using gnathodynamometer to compare the difference between maximum biting force

IPD SHARING:
Plan to Share IPD: No
data will be available through contact by email of the princible investigator ( ahmed_saad@dentistry.cu.ed.eg)

REFERENCES:
- [Background] 1. Brunello DL, Mandikos MN (1998) Construction faults, age, gender, and relative medical health: factors associated with complaints in complete denture patients. J Prosthet Dent 79, 545-554. 2. Craig RG, Powers JM, et al. Restorative Dental Materials. 11th ed. St Louis: Mo, Mosby; 2002. pp. 636-689. 3. O Bricn WJ. Dental Material and their selection. 4th ed. Chicago: Quintessence Publishing Co, Inc.; 2008. pp. 75-113. 4. Marei MK. Reinforcement of denture base resin with glass fillers. J Prosthodont. 1999; 8: 18-26. 5. Vojdani M, Khaledi AAR. Transverse Strength of Reinforced Denture Base Resin with Metal Wire and E-Glass Fibers. J Dent Tehran Univ Med Scien. 2006; 3: 167-172. 6. Vojdani M, Bagheri R, Khaledi AAR. Effects of aluminum oxide addition on the flexural strength, surface hardness, and roughness of heat-polymerized acrylic resin. Journal of Dental Sciences. 2012; 7: 238-244. 7. Matthews E, Smith DC. Nylon as a denture base material. Br Dent J. 1955; 98: 231-237. 8. Negrutiu Meda et al (2005) Thermoplastic resins for ﬂexible framework removable partial dentures. TMJ 55:3 9. Hazari, P., Bhoyar, A., Mishra, S. K., Yadav, N. S., & Mahajan, H. (2015). A Comparison of Masticatory Performance and Efficiency of Complete Dentures Made with High Impact and Flexible Resins: A Pilot Study. Journal of Clinical and Diagnostic Research : JCDR, 9(6), ZC29-34. doi:10.7860/JCDR/2015/12207.6089 10. Rueggeberg FA. From Vulcanite to vinyl, a history of resins in restorative dentistry, J Prosthet Dent. 2002; 87(4):364-79.